CLINICAL TRIAL: NCT03566303
Title: Rivaroxaban vs Warfarin in Patients With Metallic Prosthesis
Acronym: RIWA
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Coronavirus Pandemic
Sponsor: Hospital Geral Roberto Santos (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 90288318.0.0000.5028
Record Dates: First submitted 2018-06-08; First posted 2018-06-25 (Actual); Last update posted 2020-05-15 (Actual); Status verified 2020-05

CONDITIONS: Prostheses and Implants; Stroke; Valve Heart Disease; Anticoagulants and Bleeding Disorders
Keywords: Valve Heart Disease; Rivaroxaban; Warfarin
MeSH Terms: conditions — Stroke; Heart Valve Diseases; Hemostatic Disorders | interventions — Rivaroxaban; Warfarin; acarboxyprothrombin

STUDY DESIGN:
Intervention Model Description: It was adopted an equal allocation of patients to each treatment (i.e., 1:1 randomization)
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Rivaroxaban (Active Comparator): Rivaroxaban 15mg BID
  Interventions: Drug: Rivaroxaban 15 mg
- Warfarin (Placebo Comparator): Warfarin dose adjusted
  Interventions: Drug: Warfarin

INTERVENTIONS:
Drug: Rivaroxaban 15 mg — Rivaroxaban 15 mg BID
  Other Names: Xarelto 15 mg; Rivaroxabana 15 mg
  Arms: Rivaroxaban
Drug: Warfarin — Warfarin
  Other Names: Vitamin K antagonist
  Arms: Warfarin

SUMMARY:
Mechanical heart valves (MHV) demand lifelong anticoagulation with vitamin K antagonists (VKA) due to the high thrombogenicity of the prosthesis. Rivaroxaban has previously been tested in experimental and animal models with encouraging results. The investigators recently sent for publication an experiment with 7 patients who used rivaroxaban in metallic prosthesis with encouraging results. In this way it was decided to do a randomized non-inferiority clinical trial comparing rivaroxaban with warfarin in patients with metallic prosthesis.

DETAILED DESCRIPTION:
For patients with severe and symptomatic valvular heart disease, valve replacement surgery improves morbidity and mortality outcomes. It is estimated that four million valve replacement procedures have been performed over the last 50 years and it remains the only definitive treatment for most patients with advanced heart valve disease.1 Patients who received mechanical heart valves (MHV) had a significantly lower mortality, higher cumulative incidence of bleeding and, in some age groups, stroke than did recipients of a biologic prosthesis. In addition, MHV demands lifelong anticoagulation with vitamin K antagonists (VKA), most commonly warfarin, due to the high thrombogenicity of the prosthesis. Even with the appropriate use of therapy, there is a high incidence of thromboembolic events: 1% to 4% per year. Furthermore, bleeding risk is significant, ranging from 2% to 9% per year.4 Indeed, variability in the international normalized ratio (INR) is a major independent predictor of reduced survival in patients with MHV.5 Due to the narrow therapeutic index, interactions, genetic variants, and need for blood monitoring of patients taking VKAs, alternatives to warfarin have now been made available: specifically, inhibitors that directly target Factor IIa (dabigatran) or Xa (rivaroxaban, apixaban, edoxaban).6 RE-ALIGN was a prospective, randomized, phase 2, open-label trial that randomized 252 patients within a 2:1 unblinded fashion to either dabigatran or warfarin, with patients stratified according to interval since replacement (within three to seven days in population A; >three months in population B). Unfortunately, the trial was terminated prematurely because of an excess of thromboembolic and bleeding events among patients in the dabigatran group. The negative results of this study can be explained by the selection of 50 ng/mL as the target dabigatran trough level, the possibility of this drug inducing downstream effects on the coagulation cascade that impair its ability to blunt the postoperative hypercoagulable state relative to warfarin and the inclusion of early postoperative patients (population A) since it is a phase of high incidence of thromboembolic events.

On the other hand, rivaroxaban has already been tested in experimental9 and animal models10 with encouraging results. According to these findings, the investigators hypothesized that a direct Factor Xa inhibitor could be evaluated in patients with MHV for prevention of thromboembolic events.

ELIGIBILITY:
Inclusion Criteria:

- Mechanical prosthetic valve replacement after at least 3 months postoperative

Exclusion Criteria:

* Previous hemorrhagic stroke
* Ischemic stroke in the last 3 months
* Severe renal impairment (CrCl rates < 30 ml/min)
* Active liver disease (any etiology)
* Concomitant use of any antiplatelet (aspirin, clopidogrel, prasugrel, ticagrelor, ticlopidine, etc.)
* Increased risk of bleeding (congenital or acquired)
* Uncontrolled SAH
* Gastrointestinal hemorrhage within the past year
* Anemia (Hb level < 10 g/dl) or thrombocytopenia (platelet count < 100 × 109/l)
* Active infective endocarditis
* Pregnant or lactating women

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2018-07-10 (Actual); Primary Completion 2020-04-26 (Actual); Study Completion 2020-04-26 (Actual)

PRIMARY OUTCOMES:
Patients with thromboembolic events: Stroke, transient ischemic attack (TIA), silent brain infarction (SBI) and systemic embolism (SE). | 90 days
  The primary endpoint was defined as stroke, TIA, SBI and systemic embolism
major or clinically relevant nonmajor bleeding | 90 days
  The primary safety outcome was major or clinically relevant nonmajor bleeding according to the International Society on Thrombosis and Haemostasis (ISTH) criteria and Bleeding Academic Research Consortium (BARC)

SECONDARY OUTCOMES:
Patients with e of stroke/TIA/SBI/SE and/or death from any cause. | 90 days
  Combined outcome
Cases of myocardial infarction during of follow-up | 90 days
  Myocardial infarction in the course of treatment
New cases of valve thrombosis with or without symptoms | 90 days
  Clinical or asymptomatic valve thrombosis
New intracardiac thrombus detected at the end of clinical follow-up by transesophageal echocardiogram | 90 days
  Emergence of intracardiac thrombus seen on transesophageal echocardiogram

OTHER OUTCOMES:
Cases of minor bleeding | 90 days
  Any minor bleeding

CONTACTS AND LOCATIONS:
Overall Officials: Andre Duraes, PhD, Principal Investigator — Federal University of Bahia
Locations (1):
- Andre Duraes, Salvador, Estado de Bahia, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Duraes AR, de Souza Lima Bitar Y, Schonhofen IS, Travassos KSO, Pereira LV, Filho JAL, Neto MG, Junior RA, Roever L. Rivaroxaban Versus Warfarin in Patients with Mechanical Heart Valves: Open-Label, Proof-of-Concept trial-The RIWA study. Am J Cardiovasc Drugs. 2021 May;21(3):363-371. doi: 10.1007/s40256-020-00449-3. Epub 2020 Nov 5. PMID 33150497
- [Derived] Duraes AR, de Souza Lima Bitar Y, Filho JAL, Schonhofen IS, Camara EJN, Roever L, Cardoso HEDP, Akrami KM. Rivaroxaban versus Warfarin in Patients with Mechanical Heart Valve: Rationale and Design of the RIWA Study. Drugs R D. 2018 Dec;18(4):303-308. doi: 10.1007/s40268-018-0249-5. PMID 30293126